CLINICAL TRIAL: NCT06536335
Title: Evaluation of the Perceived Experience of Patients Treated With Aligners With Two Different Attachment Placement Times: Randomised Controlled Clinical Trial
Brief Title: Evaluation of the Perceived Experience of Patients Treated With Aligners With Two Different Timings
Acronym: ALLIN-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6636
Record Dates: First submitted 2024-07-18; First posted 2024-08-02 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Malocclusion
Keywords: Attachment; Discomfort; Malocclusion; Questionnaires
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: The investigator does not know to which group the patient who sent in the questionnaire belongs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional protocol (Active Comparator): A group of patients a group of patients to whom attachments will be bonded at the beginning of the first aligner.
  Interventions: Device: Biomax Nuvola aligners
- Delayed protocol (Experimental): A group of patients to whom attachments will be bonded at the beginning of the third aligner, approximately one month after the start of orthodontic treatment.
  Interventions: Device: Biomax Nuvola aligners

INTERVENTIONS:
Device: Biomax Nuvola aligners — All patients will be treated with Biomax Nuvola aligners built based on the individual patient's characteristics. The number of aligners and the number/type of attachments will be chosen on the basis of the individual malocclusions. In this group the attachments will be bonded at the beginning of first aligner. Two different questionnaires will be administered to the enrolled subjects: the italian version of the adapted OHIP-14 questionnaire, and a customized questionnaire. The questionnaires will be completed at different stages of orthodontic treatment, as following: 24 hours after the delivery of the first aligner - start of orthodontic treatment; 3 days after the start of orthodontic treatment; 7 days after the start of orthodontic treatment; 24 hours after delivery of the third clear aligner; 3 days after delivery of the third clear aligner; 7 days after delivery of the third clear aligner.
  Arms: Conventional protocol
Device: Biomax Nuvola aligners — All patients will be treated with Biomax Nuvola aligners built based on the individual atient's characteristics. The number of aligners and the number/type of attachments will be chosen on the basis of the individual malocclusions. In this group the attachments will be bonded at the beginning of third aligner, approximately one month after the start of orthodontic treatment. Two different questionnaires will be administered to the enrolled subjects: the italian version of the adapted OHIP-14 questionnaire, and a customized questionnaire. The questionnaires will be completed at different stages of orthodontic treatment, as following: 24 hours after the delivery of the first aligner - start of orthodontic treatment; 3 days after the start of orthodontic treatment; 7 days after the start of orthodontic treatment; 24 hours after delivery of the third clear aligner; 3 days after delivery of the third clear aligner; 7 days after delivery of the third clear aligner.
  Arms: Delayed protocol

SUMMARY:
The primary aim of the study is to compare the perception of pain and discomfort with two different protocols of attachments' placement during clear aligner therapy: the conventional protocol (CP), when attachments' placement is performed are placed at the delivery of the first aligner; the delayed protocol (DP), when the attachments' placement is performed at the delivery of the third aligner. The rationale of this study is to evaluate whether dividing the two phases most associated with the onset of pain and discomfort, namely the initiation of aligner therapy and the placement of attachments, can improve patients' quality of life during clear aligner treatment. Patients' discomfort will be evaluated with a questionnaire adapted by OHIP-14 (Oral Health Impact Profile 14)

DETAILED DESCRIPTION:
: The study was approved by the Institutional Review board of the Catholic University of the Sacred Hearth, Rome, Italy (prot. n. 17048/23). All adult patients with class I and II malocclusion referred to the Fondazione Policlinico Universitario Agostino Gemelli will be consecutively enrolled for this study. All patients will be treated with Biomax Nuvola aligners built based on the individual patient's characteristics. The number of aligners and the number/ type of attachments will be chosen on the basis of the individual malocclusions.

Patients will be randomly allocated in two different groups: the study group includes patients following the delayed protocol (DP), while the control group is composed of patients' following the conventional protocol (CP). The aligner will be changed every 15 days, so the attachment placement in the DP will be performed around 30 days from the beginning of the clear aligner treatment. The modified OHIP Italian version has 20 questions categorized into 7 sections, concerning the limitation generated by deterioration of oral health in relation to clear aligners: functional, pain, psychological discomfort, physical or psychological or social disability, and handicap. The answers range from 0 (never) to 4 (very often). Possible categories are: never (0), rarely (1), sometimes (2), habitually (3), and very often (4). Low scores indicate better self-perception of quality of life. The customised questionnaire has 9 questions, concerning the limitation generated by discomfort caused by attachments. For 8 questions, the answers range from 0 (never) to 4 (very often). Possible categories are: never (0), rarely (1), sometimes (2), habitually (3), and very often (4). Low scores indicate better self-perception of quality of life. For the last question the answer is based on NRS scale, in fact it ranges from 0 to 10. Lower score indicates less pain perceived by the patient. The questionnaires will be filled out at different phases of orthodontic treatment, specifically: at the delivery of the first aligner, after 3 and 7 days; at the delivery of the third aligner, after 3 and 7 days. The survey scheduling is arranged according to White, who stated that the patients' perception of pain and discomfort occurred within 7 days after the beginning of the orthodontic treatment; then, patients' quality of life tends to return to a baseline condition.

The study will be single-blind, because the person collecting the results and making the assessments will not know which treatment was used. In fact, the patient will anonymously submit the answers to the questionnaires uploaded on Microsoft Form, using an acronym that will be provided to him/her by the clinical operator. In this way, the person collecting and analysing the data will not know to which group the patient who sent the answers belongs.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years;
* Class I malocclusion
* Non-extractive treatment;
* No missing teeth (third molars excluded);
* Good oral and general health.
* Signature of written informed consent to participate in the study

Exclusion Criteria:

* Patients with tooth-related pain (presence of dental and/or periodontal abscesses and presence of gingivitis)
* Presence of semi-included elements;
* Patients taking bisphosphonates or other anti-resorptive drugs;
* Patients with conditions involving chronic pain and/or on chronic therapy with antifiammatories/opiods or other drugs that may act on pain perception;
* Patients with temporomandibular disorders;
* Patients with conditions that may impair the ability to objectively report any sensations of discomfort or pain (e.g., mental retardation, dementia);
* Refusal to sign the written informed consent to participate in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of a possible reduction in discomfort between the two protocols | 1 year
  The primary objective of the study is to evaluate whether splitting the two phases most associated with the onset of pain and discomfort,i.e. the initiation of aligner therapy and the placement of attachments,can reduce these sensations and, consequently,improve adherence to treatment.Specifically,the level of pain symptomatology perceived by the patient will be assessed using the OHIP-14 scale.
  The OHIP version has 14 questions,concerning the limitation generated by oral health impairment:functional limitation, pain, psychological discomfort, physical disability, psychological disability,social disability, and disability. The possible answers are: never (0), rarely (1), sometimes (2), habitually (3), and very often (4). The score is given by the sum of the values,from a minimum of 0 points to a maximum of 56 points.

SECONDARY OUTCOMES:
Different timing of onset and disappearance of pain | 1 year
  Evaluation of whether the two protocols are associated with different timing of onset and disappearance of pain. In particular, this issue will be evaluated using a questionnaire developed for the study, with questions concerning the presence of discomfort due to aligner treatment and resin composite attachment. This questionnaire has 8 questions and the possible answers are: never(0), rarely(1), sometimes(2), habitually(3), and very often(4). The score is given by the sum of the values from a minimum of 0 points to a maximum of 32.This questionnaire will be sent with different timing, specifically:
  * 24 hours after the start of orthodontic treatment;
  * 3 days after the start of orthodontic treatment;
  * 7 days after the start of orthodontic treatment;
  * 24 hours after delivery of the third aligner;
  * 3 days after delivery of the third aligner;
  * 7 days after delivery of the third aligner.
Impact on patients' quality of life | 1 year
  Evaluate if the two protocols impact patients' quality of life differently. Specifically, the extent of pain symptomatology perceived by the patient will be assessed by the masked operator using the NRS scale (score 0-10, the lower it is, the less pain is perceived by the patient).

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cordaro, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC odontoiatria, Roma, Italy

REFERENCES:
- [Background] Weir T. Clear aligners in orthodontic treatment. Aust Dent J. 2017 Mar;62 Suppl 1:58-62. doi: 10.1111/adj.12480. PMID 28297094
- [Background] Bergius M, Kiliaridis S, Berggren U. Pain in orthodontics. A review and discussion of the literature. J Orofac Orthop. 2000;61(2):125-37. doi: 10.1007/BF01300354. English, German. PMID 10783564
- [Background] Bergius M, Berggren U, Kiliaridis S. Experience of pain during an orthodontic procedure. Eur J Oral Sci. 2002 Apr;110(2):92-8. doi: 10.1034/j.1600-0722.2002.11193.x. PMID 12013568
- [Background] Rakhshan H, Rakhshan V. Pain and discomfort perceived during the initial stage of active fixed orthodontic treatment. Saudi Dent J. 2015 Apr;27(2):81-7. doi: 10.1016/j.sdentj.2014.11.002. Epub 2015 Jan 27. PMID 26082574
- [Background] Lew KK. Attitudes and perceptions of adults towards orthodontic treatment in an Asian community. Community Dent Oral Epidemiol. 1993 Feb;21(1):31-5. doi: 10.1111/j.1600-0528.1993.tb00715.x. PMID 8432102
- [Background] Antonio-Zancajo L, Montero J, Albaladejo A, Oteo-Calatayud MD, Alvarado-Lorenzo A. Pain and Oral-Health-Related Quality of Life in Orthodontic Patients During Initial Therapy with Conventional, Low-Friction, and Lingual Brackets and Aligners (Invisalign): A Prospective Clinical Study. J Clin Med. 2020 Jul 3;9(7):2088. doi: 10.3390/jcm9072088. PMID 32635196
- [Background] Tamer I, Oztas E, Marsan G. Orthodontic Treatment with Clear Aligners and The Scientific Reality Behind Their Marketing: A Literature Review. Turk J Orthod. 2019 Dec 1;32(4):241-246. doi: 10.5152/TurkJOrthod.2019.18083. eCollection 2019 Dec. PMID 32110470
- [Background] White DW, Julien KC, Jacob H, Campbell PM, Buschang PH. Discomfort associated with Invisalign and traditional brackets: A randomized, prospective trial. Angle Orthod. 2017 Nov;87(6):801-808. doi: 10.2319/091416-687.1. Epub 2017 Jul 28. PMID 28753032
- [Background] Cardoso PC, Espinosa DG, Mecenas P, Flores-Mir C, Normando D. Pain level between clear aligners and fixed appliances: a systematic review. Prog Orthod. 2020 Jan 20;21(1):3. doi: 10.1186/s40510-019-0303-z. PMID 31956934
- [Background] Almasoud NN. Pain perception among patients treated with passive self-ligating fixed appliances and Invisalign(R) aligners during the first week of orthodontic treatment. Korean J Orthod. 2018 Sep;48(5):326-332. doi: 10.4041/kjod.2018.48.5.326. Epub 2018 Aug 8. PMID 30206531
- [Background] Franchignoni M, Giordano A, Brigatti E, Migliario M, Levrini L, Ferriero G. [Psychometric properties of the Italian version of the reduced form of the Oral Health Impact Profile (OHIP-14)]. G Ital Med Lav Ergon. 2010 Jul-Sep;32(3 Suppl B):B71-8. Italian. PMID 21302527
- [Background] Thong ISK, Jensen MP, Miro J, Tan G. The validity of pain intensity measures: what do the NRS, VAS, VRS, and FPS-R measure? Scand J Pain. 2018 Jan 26;18(1):99-107. doi: 10.1515/sjpain-2018-0012. PMID 29794282